CLINICAL TRIAL: NCT00578552
Title: Gabapentin for Smoking Abstinence
Brief Title: Gabapentin for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Amit Sood, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-005262; 07-000700
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2010-12-01 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Cigarette Smoking; Tobacco Use
Keywords: tobacco; smoking; gabapentin; abstinence
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use; Smoking | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Non active placebo pill
  Interventions: Drug: Placebo
- Gabapentin - 1800 mg/day (Active Comparator): Gabapentin - 1800 mg/day
  Interventions: Drug: Gabapentin - 1800 mg/day
- Gabapentin - 2700 mg/day (Active Comparator): Gabapentin - 2700 mg/day
  Interventions: Drug: Gabapentin - 2700 mg/day

INTERVENTIONS:
Drug: Placebo — Placebo pill - non active sugar pill designed to look alike to the gabapentin medication
  Arms: Placebo
Drug: Gabapentin - 1800 mg/day — gabapentin - 1800 mg/day for 12 weeks.
  Other Names: gabapentin
  Arms: Gabapentin - 1800 mg/day
Drug: Gabapentin - 2700 mg/day — gabapentin - 2700 mg/day for 12 weeks.
  Other Names: gabapentin
  Arms: Gabapentin - 2700 mg/day

SUMMARY:
Gabapentin is an anti-epileptic agent that has shown preliminary evidence of efficacy for improving symptoms of cocaine and alcohol withdrawal in pilot studies. Since the neurobiology of alcohol, cocaine and nicotine withdrawal is similar, the preliminary evidence of efficacy of gabapentin for symptoms of alcohol and cocaine withdrawal suggests, that gabapentin might likely help nicotine withdrawal symptoms and thus tobacco abstinence. The effect of gabapentin on two of the neurotransmitters, gamma-aminobutyric acid (GABA) and glutamate further suggest a potential therapeutic mechanism for gabapentin in tobacco abstinence. However, the exact mechanism of action of gabapentin is currently not known. We have recently completed an open label pilot trial of gabapentin for tobacco abstinence involving 50 smokers. The findings from that study provide promising preliminary results and suggest that further testing of gabapentin for helping cigarette smokers quit tobacco use is worth pursuing. Overall, gabapentin is well tolerated and has low abuse potential.

Our goal is to evaluate novel, safe, acceptable, and effective therapies that may help increase tobacco abstinence rates. Currently, no randomized trials testing the efficacy of gabapentin for smoking abstinence have been published. While our previous study provides promising evidence regarding the potential efficacy of gabapentin for smoking abstinence, an additional dose ranging study is needed prior to pursuing a large randomized trial. The primary aim of the dose ranging study will be to obtain additional evidence of efficacy, and information on the optimal dose of gabapentin to employ in the larger randomized controlled trial.

DETAILED DESCRIPTION:
A total of 120 participants will be recruited in this study and randomly assigned to one of the three groups. Participants in group A will receive gabapentin 1800-mg/day orally for 12-weeks while participants in group B will receive gabapentin 2700-mg/day orally for 12-weeks. Participants in group C will receive a matching placebo for the same duration. We have selected this dose regimen based on our experience with using gabapentin in the pilot study. The present study is designed as a randomized, blinded, placebo-controlled, three-arm, parallel-group, dose-ranging, phase II clinical trial. In addition to receiving gabapentin or placebo, all subjects will receive a brief behavioral counseling intervention during participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Are between 18 to 65 years of age
2. Have smoked ≥10 cigarettes/day for the past 1 year or more
3. Are willing to make a quit attempt
4. Are able to participate fully in all aspects of the study; and
5. Have been provided with, understand, and have signed the informed consent.

Exclusion Criteria:

1. Meet diagnostic criteria for current major depressive disorder or lifetime history of bipolar disorder or schizophrenia. Patients with mild or moderate depressive symptoms as assessed by the CES-D and determined by the physician, but who do not meet current diagnostic criteria for major depressive disorder, will be included
2. Are currently (within past 30 days) using antipsychotics, or antidepressants
3. Are currently (in previous 30 days) using any tobacco treatment program (i.e., behavioral therapy, nicotine replacement therapy, bupropion SR, clonidine, or nortriptyline)
4. Have used an investigational drug within the 30 days prior to enrolling in this study
5. Have recent history (in the past year) of alcohol abuse or dependence as assessed by the CAGE questionnaire and study investigators
6. Have a recent history of drug abuse as assessed by the Drug Abuse Screening Test 20 (DAST-20) and physician interview
7. Are pregnant, lactating, or of child bearing potential, likely to become pregnant during the medication phase and not willing to use contraception. The following birth control measures are acceptable: birth control pills, approved intra-uterine contraceptive devices, the use of two combined barrier methods (diaphragm with spermicide or condom with spermicide), injections, surgical sterilization and abstinence
8. Have a history of any major cardio-vascular events in the past 6 months including unstable angina, acute MI or coronary angioplasty
9. Have clinically significant acute or chronic progressive or unstable neurologic (myasthenia gravis), hepatic, renal, cardiovascular, respiratory (bronchospastic disease) or metabolic disease
10. Are currently on the following prescribed medications known to interact with gabapentin and unable to stop them during the study: Maalox®, cimetidine and morphine. Patients will be cautioned not to use sedatives (such as benzodiazepines, antihistamines, anti-cholinergics, trazodone, zaleplon, anti-psychotics, barbiturates, opiates, zolpidem and eszopiclone) during the study
11. Have another house-hold member or relative participating in the study
12. Have known allergy to gabapentin or its constituents; and
13. Are professional drivers or operators of heavy machinery and unable to refrain from these activities during the medication phase of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sood, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Nicotine Research Program, Rochester, Minnesota, United States

REFERENCES:
- [Result] Sood A, Ebbert JO, Wyatt KD, Croghan IT, Schroeder DR, Sood R, Hays JT. Gabapentin for smoking cessation. Nicotine Tob Res. 2010 Mar;12(3):300-4. doi: 10.1093/ntr/ntp195. Epub 2010 Jan 15. PMID 20081039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 08/07/2007 and completed on 12/10/2008. Interested subjects who passed a phone pre-screen were seen at a medical clinic (Mayo Clinic in Rochester, MN and Franciscan Skemp Medical Center in Lacrosse, WI) for consenting and additional study procedures to determine eligibility.
Groups:
- Placebo: Placebo pill was identical in appearance to the active medication. Initial dosage consisted of 1 pill by mouth in the morning and night. The dose was increased over the first 2 weeks to the target frequency of three times a day. This dose was continued for the next 9 weeks and tapered in the last week. The medication was stopped at the end of 12 weeks.
- Gabapentin - 1800 mg /Day: Gabapentin was initiated at a dose of 300 mg by mouth in the morning and night. The dose was increased over the first 2 weeks to the target doses of 600 mg three times a day. This dose was continued for the next 9 weeks and tapered in the last week. The medication was stopped at the end of 12 weeks.
- Gabapentin - 2700 mg/Day: Gabapentin was initiated at a dose of 300 mg by mouth in the morning and night. The dose was increased over the first 2 weeks to the target doses of 900 mg three times a day. This dose was continued for the next 9 weeks and tapered in the last week. The medication was stopped at the end of 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Gabapentin - 1800 mg /Day | Gabapentin - 2700 mg/Day
Started | 27 | 27 | 26
Completed | 12 | 13 | 11
Not Completed | 15 | 14 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Gabapentin - 1800 mg /Day | Gabapentin - 2700 mg/Day | Total
Number analyzed (Participants) | 27 | 27 | 26 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 26 | 80
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.0 (11.1) | 41.1 (9.5) | 40.7 (13.5) | 40.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 8 | 30
  Male | 16 | 16 | 18 | 50
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] — Self Reported average number of cigarettes smoked per day in the preceeding 6 months prior to study enrollment.
  cigarettes per day | 20.0 (6.6) | 23.7 (6.9) | 20.9 (7.9) | 21.5 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Biochemically Confirmed 7-day Point Prevalence Abstinence From Tobacco
Description: Point prevalence tobacco abstinence was adjudicated if the following conditions were met: (a) self-reported tobacco abstinence for the previous 7 days with a negative response to the question "Have you used any type of tobacco, even a puff, in the past 7 days?" and (b) Expired Carbon Monoxide equal or less then 8 parts per million.
Time Frame: 12 weeks following start of medication
Measure: Number; unit: participants
Arm/Group | Placebo | Gabapentin - 1800 mg /Day | Gabapentin - 2700 mg/Day
Number analyzed (Participants) | 27 | 27 | 26
participants | 5 | 4 | 0
Statistical Analysis 1: Comparison: Placebo vs Gabapentin - 1800 mg /Day; Data were compared between treatment groups using Fisher's exact test for binary outcomes; Test type: Superiority or Other; p = 0.77, Fisher Exact; 1-tailed
Statistical Analysis 2: Comparison: Placebo vs Gabapentin - 2700 mg/Day; Data were compared between treatment groups using Fisher's exact test for binary outcomes; Test type: Superiority or Other; p = 1.00, Fisher Exact; 1-tailed

ADVERSE EVENTS:
Time Frame: All adverse events were collected for the duration of the treatment phase (up to 12 weeks following start of medication). SERIOUS adverse events were collected for the duration of the study (6 months).
Arm/Group | Placebo | Gabapentin - 1800 mg /Day | Gabapentin - 2700 mg/Day
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/27 | 1/26
Other Adverse Events (participants affected / at risk) | 5/27 | 12/27 | 7/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | Gabapentin - 1800 mg /Day (N=27) | Gabapentin - 2700 mg/Day (N=26)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 — Study participant reported having a Heart Attack during the follow up phase of the study (post medication phase). This was determined NOT to be related to the study drug.
Alcohol Intoxication (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Subject became intoxicated and had to be hospitalized while in the study medication phase of the study. The attending physician and PI did not determine this to be related to study medication.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | Gabapentin - 1800 mg /Day (N=27) | Gabapentin - 2700 mg/Day (N=26)
Dizziness (General disorders) | 1 | 4 | 4
Decreased Concentration (General disorders) | 0 | 3 | 0
Edema (General disorders) | 1 | 2 | 0
Sleep Disturbance (General disorders) | 3 | 0 | 0
Ataxia (General disorders) | 0 | 1 | 1
Dry Mouth (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 0 | 2 | 0
Headache (General disorders) | 1 | 1 | 0
Nausea (General disorders) | 1 | 1 | 0
Rash (General disorders) | 0 | 1 | 1
Hand Tremors (General disorders) | 0 | 0 | 1
Increased Energy (General disorders) | 0 | 1 | 0
Polyuria (General disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The original intent was to enroll a total of 120 subjects. However, due to the high study dropout rate, a review of the primary endpoint was performed after 80 subjects were enrolled and a decision was made to discontinue further enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes